CLINICAL TRIAL: NCT05000346
Title: A Randomized, Double-blind, Placebo-controlled, Parallel, Trial to Determine the Safety and Efficacy of Inhaled AQ001S in the Management of Acute COVID-19 Symptoms
Brief Title: Clinical Trial to Assess the Efficacy and Safety of Inhaled AQ001S in the Management of Acute COVID-19 Symptoms
Acronym: SIROCCO-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of patient to recruit
Sponsor: Aquilon Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AQ-PRO-013
Record Dates: First submitted 2021-06-24; First posted 2021-08-11 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Pharmaceutical Preparations; Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental AQ001S 0.125 mg/mL quarter in die (Experimental): AQ001S 0.125 mg/mL inhalation solution administered by inhalation 4 times a day
  Interventions: Drug: Drug, inhalation
- Experimental AQ001S 0.125 mg/mL bis in die (Experimental): AQ001S 0.125 mg/mL inhalation solution administered by inhalation twice a day + placebo by inhalation twice a day
  Interventions: Drug: Drug, inhalation
- Comparator: placebo (Placebo Comparator): No active drug - administered by inhalation 4 times a day
  Interventions: Drug: Drug, inhalation

INTERVENTIONS:
Drug: Drug, inhalation — Solution administered by inhalation
  Other Names: inhaled drug, including placebo

SUMMARY:
Double-blind parallel trial to assess the efficacy and safety of inhaled AQ001S in the management of acute COVID-19 symptoms compared.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, parallel clinical trial to determine the safety and efficacy of inhaled AQ001S in the management of acute COVID-19 symptoms in adult patients (≥ 18 years old) who are admitted to hospital due to the severity of his/her confirmed or suspected COVID-19 disease. The patient will be treated for 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Patient admitted to hospital due to the severity of his/her confirmed or suspected COVID-19 disease.
2. Positive virus test for Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) using real time polymerase chain reaction (nasal swab).
3. Patient with COVID-19 clinical progression scale score ≥ 4 (hospitalized; no oxygen therapy).
4. Male or female, ≥18 years of age at the time of consent.
5. Patients who have given written informed consent.
6. Reliable patients who are willing to be available for the duration of the clinical trial and willing to comply with clinical trial procedures.
7. Patients who have the ability to understand the requirements of the clinical trial.
8. Female patients of childbearing potential (women of childbearing potential, WOCBP ) should have a negative pregnancy test at Screening Visit.
9. Female patients of childbearing potential (women of childbearing potential, WOCBP1) using a highly effective method of contraception (i.e., pregnancy rate of < 1% per year) on a stable regimen, for at least 28 days, and pursuing this contraception during the trial and for 28 days after the last administration of the study drug The highly effective methods of contraception must be one of the following: combined estrogen and progestogen hormonal contraception with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner, or agreement on continuous abstinence from heterosexual intercourse.

Exclusion Criteria:

1. Intensive care patients
2. Inability to use a nebulizer with a mouthpiece.
3. History of hypersensitivity to corticosteroid or to any of the excipients in the drug preparation.
4. Untreated oral candidiasis.
5. Evidence of symptomatic chronic or acute respiratory infection other than COVID-19 in the previous 8 weeks.
6. Proven diagnosis of Chronic Obstructive Pulmonary Disease, asthma or bronchiectasis.
7. Pulmonary malformations, tuberculosis, cystic fibrosis.
8. History or presence of severe renal (stage 4 (GFR = 15-29 mL/min)) and/or severe hepatic impairment(s) (grade 4 or above)
9. Anticipated transfer to another hospital within 72 hours.
10. Use of inhaled corticosteroid, at a strength at least equivalent to 200 µg of beclomethasone per day, within 7 days before Screening Visit.
11. Systemic corticosteroids (e.g., dexamethasone) within 28 days before Screening Visit.
12. Female patients who are breast-feeding, lactating, pregnant or intending to become pregnant.
13. Any condition, including findings in the patients' medical history or in the pre-randomization study assessments that, in the opinion of the Investigator, constitute a risk or a contraindication for the participation of the patient into the study or that could interfere with the study objectives, conduct or evaluation.
14. Current or previous participation in another clinical trial where the patient has received a dose of an study drug containing small molecules within 30 days or 5 half-lives (whichever is longer) prior to entry into this study or containing biologicals within 3 months prior to entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | During 28 days of treatment
  Incidence of Treatment-Emergent Adverse Events as assessed by collection of (Serious) Adverse Events and general/local tolerability
WHO clinical progression scale (COVID-19 clinical progression scale) | At Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2 (Visit 5)
  Change in the WHO clinical progression scale (reference: WHO Working Group on the Clinical Characterisation and Management of COVID-19 infection, Lancet Infect Dis., Aug 2020, 20(8): e192-e197) with "Uninfected" as minimal value (e.g. 0) and "Dead" as maximal value (e.g. 10, worse outcome), ffrom baseline (Visit 2) to Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2.

SECONDARY OUTCOMES:
Time to hospital discharge | After 28 days of treatment
  Time to hospital ldischarge measured over the treatment period from baseline (visit 2) to day 28 (visit 5).
Time to Intensive Care Unit admission | After 28 days of treatment
  Time to Intensive Care Unit admission measured over the treatment period from baseline (visit 2) to day 28 (visit 5).
Length of Intensive Care Unit stay | After 28 days of treatment
  Length of Intensive Care Unit stay measured over the treatment period from baseline (visit 2) to day 28 (visit 5).
Time to hospital readmission | After 28 days of treatment
  Time to hospital readmission measured over the treatment period from baseline (visit 2) to day 28 (visit 5).
Length of hospital readmission | After 28 days of treatment
  Length of hospital readmission measured over the treatment period from baseline (visit 2) to day 28 (visit 5).
Time to mechanical ventilation | After 28 days of treatment
  Time to mechanical ventilation measured over the treatment period from baseline (visit 2) to day 28 (visit 5).
Occurrence of death | Within 60 days from hospitalisation
  Occurence of death (all deaths).
Modified Medical Research Council Dyspnea Scale | to Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2 (Visit 5)
  Change in modified Medical Research Council Dyspnea (mMRC) Scale from baseline (Visit 2) to Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2 (Visit 5).
  Minimum mMRC Scale value is 0 (e.g. "I only get breathless with strenuous exercise"). The maximum mMRC Scale value is 4 (e.g. "I am too breathless to leave the house" or "I am breathless when dressing", worse outcome).
Pulmonary function measurement: Forced Expiratory Volume in the first second (FEV1) | At Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2 (Visit 5)
  Changes in FEV1 measured from baseline (Visit 2) to Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2.
Pulmonary function measurement: Forced Vital Capacity (FVC) | At Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2 (Visit 5)
  Changes in FVC measured from baseline (Visit 2) to Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2.
Pulmonary function measurement: FEV1/FVC ratio | At Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2 (Visit 5)
  Changes in FEV1/FVC ratio from baseline (Visit 2) to Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2.
Pulmonary function measurement: Oxygen saturation (SpO2) | At Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2 (Visit 5)
  Changes in SpO2 measured from baseline (Visit 2) to Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2.
Pulmonary function measurement: Fraction of inspired Oxygen (FiO2) | At Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2 (Visit 5)
  Changes in FiO2 measured from baseline (Visit 2) to Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2.
Pulmonary function measurement: SpO2/FiO2 ratio | At Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2 (Visit 5)
  Changes in and SpO2/FiO2 ratio measured from baseline (Visit 2) to Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2.
Diffusion Capacity for Carbon Monoxide measurements | At Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2 (Visit 5)
  Changes in the Diffusion Capacity for Carbon Monoxide (DLCO) from baseline (Visit 2) to Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2.
Pulmonary CT Scan | After 28 days of treatment
  Changes in the pulmonary CT Scan between baseline (Visit 2) and Day 28±2 (Visit 5)

OTHER OUTCOMES:
Change immune system response | After 28 days of treatment
  Changes in the immune system response will be measured from baseline (Visit 2) to Day 28±2 (Visit 5), using a 15-plex Human Cytokine Panel assay.
Change in monocyte count | After 28 days of treatment
  Changes in monocyte count will be measured from baseline (Visit 2) to Day 28±2 (Visit 5).
Change in lymphocyte count | After 28 days of treatment
  Changes in lymphocyte count will be measured from baseline (Visit 2) to Day 28±2 (Visit 5).
Change in hyperinflammation biomarker: ferritin | After 28 days of treatment
  Changes in hyperinflammation biomarkers will be measured from baseline (Visit 2) to Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2.
Change in hyperinflammation biomarker: C reactive protein | After 28 days of treatment
  Changes in hyperinflammation biomarkers will be measured from baseline (Visit 2) to Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2.
Change in hyperinflammation biomarker: d-dimer | After 28 days of treatment
  Changes in hyperinflammation biomarkers will be measured from baseline (Visit 2) to Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2.
Change in hyperinflammation biomarker: soluble cluster of differentiation 40 ligand | After 28 days of treatment
  Changes in hyperinflammation biomarkers will be measured from baseline (Visit 2) to Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2.
Change in hyperinflammation biomarker: matrix metalloproteinase | After 28 days of treatment
  Changes in hyperinflammation biomarkers will be measured from baseline (Visit 2) to Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2.
Change in cardiovascular biomarker: troponin | After 28 days of treatment
  Changes in troponin level will be measured from baseline (Visit 2) to Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2.
Change in cardiovascular biomarker: creatine kinase | After 28 days of treatment
  Changes increatine kinase level will be measured from baseline (Visit 2) to Day 7±2 (Visit 3), Day 14±2 (Visit 4) and Day 28±2.
Immunology parameters: immunoglobulin E | After 28 days of treatment
  Changes in immunoglobulin E rates from baseline (Visit 2) to Day 28±2 (Visit 5), and at each visit over the dosing period
Immunology parameters: immunoglobulin A | After 28 days of treatment
  Changes in immunoglobulin A rates from baseline (Visit 2) to Day 28±2 (Visit 5), and at each visit over the dosing period
Immunology parameters: immunoglobulin G | After 28 days of treatment
  Changes in immunoglobulin G rates from baseline (Visit 2) to Day 28±2 (Visit 5), and at each visit over the dosing period

CONTACTS AND LOCATIONS:
Overall Officials: Julien Guiot, MD, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (1):
- CHU Liege, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No